CLINICAL TRIAL: NCT02416947
Title: The Effect of Soluble Corn Fiber (SCF) on Bone Resorption in Post-Menopausal Women Using 41Calcium Technology
Brief Title: Soluble Corn Fiber Effect on Bone Resorption in Post Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Tate & Lyle Health & Nutrition Sciences (Unknown)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: TateLyle Ca41
Record Dates: First submitted 2015-04-08; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Soluble Corn Fiber; Osteoporosis; Bone Loss
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0g SCF (Placebo Comparator): Subjects will consume 0 g of SCF in two equal doses as a muffin and a drink, daily for 50 days.
  Interventions: Dietary Supplement: 0 g SCF
- 10 g SCF (Active Comparator): Subjects will consume 10 g of SCF in two equal doses as a muffin and a drink, daily for 50 days.
  Interventions: Dietary Supplement: 10g SCF
- 20g SCF (Active Comparator): Subjects will consume 20 g of SCF in two equal doses as a muffin and a drink, daily for 50 days.
  Interventions: Dietary Supplement: 20g SCF

INTERVENTIONS:
Dietary Supplement: 0 g SCF — 0 grams of SCF will be administered daily in two equal doses in the form of a muffin and a drink.
  Other Names: 0 g Soluble Corn Fiber
  Arms: 0g SCF
Dietary Supplement: 10g SCF — 10 grams of SCF will be administered daily in two equal doses in the form of a muffin and a drink.
  Other Names: 10 g Soluble Corn Fiber
  Arms: 10 g SCF
Dietary Supplement: 20g SCF — 20 grams of SCF will be administered daily in two equal doses in the form of a muffin and a drink.
  Other Names: 20 g Soluble Corn Fiber
  Arms: 20g SCF

SUMMARY:
This study is designed to study the dose response effect of continuous Soluble Corn Fiber (SCF) intake over a 50 day period on bone resorption in healthy post menopausal women using the 41Calcium methodology. To further understand the dose response effect of SCF bone biomarkers will be studied.

Our hypothesis is that soluble corn fiber will reduce bone resorption in a dose dependent manner in comparison to placebo when estimated by urinary 41Calcium excretion as well as bone biomarkers of resorption.

DETAILED DESCRIPTION:
Subjects will be dosed with 41Calcium , a long-lived radio isotope, which will become deposited in the skeleton after about 100 days. During this time subjects will collect 24 h urine monthly to monitor the decrease in 41Calcium urinary excretion. Subsequently, the baseline level of 41Calcium urinary excretion will be evaluated over a 50 day baseline period with 24 h urine collections every 10 days. Participants will then be randomized to one of three doses of soluble corn fiber (0,10,20 g/d) to be consumed in two equivalent doses per day for 50 days. Women will collect 24 h urine every 10 days. Each 50 day period will be followed by a 50 day washout period during which the subjects will continue to collect urine every 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 4 years Postmenopausal

Exclusion Criteria:

* Medications affecting bone resorption

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in 41Ca/Ca ratio in five 24 h urine collections during intervention periods compared to urinary 41Ca/Ca ratios during non-intervention periods | 24 h urine collections on days 10, 20, 30, 40, and 50 of each of three intervention periods and 4 non intervention periods
  41Ca/Ca ratio will be determined by Accelerator Mass Spectrometry. A linear regression model including the data from the non-intervention ratios will determine the predicted 41Ca/Ca ratios over the course of the 350 day study. The percent change of 41Ca/Ca ratios in the 50 day intervention periods from the predicted values will determine the effect of the intervention.

SECONDARY OUTCOMES:
Fasting serum bone specific alkaline phosphatase (BSAP), a biochemical bone formation marker | Fasting serum drawn at the end of each 50 day intervention period
Fasting serum osteocalcin (OC), a biochemical bone turnover marker | Fasting serum drawn at the end of each 50 day intervention period
Fasting urine N-terminal telopeptide, a biochemical bone resorption marker | Fasting urine collected at the end of each 50 day intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, Ph.D, Principal Investigator — Purdue University

REFERENCES:
- [Derived] Jakeman SA, Henry CN, Martin BR, McCabe GP, McCabe LD, Jackson GS, Peacock M, Weaver CM. Soluble corn fiber increases bone calcium retention in postmenopausal women in a dose-dependent manner: a randomized crossover trial. Am J Clin Nutr. 2016 Sep;104(3):837-43. doi: 10.3945/ajcn.116.132761. Epub 2016 Jul 27. PMID 27465372